CLINICAL TRIAL: NCT02657967
Title: Development of an Evidenced-Based Tool for Prediction of Sudden Death in Patients With Non-Ischemic Cardiomyopathy (NICM-Registry)
Brief Title: Development of an Evidenced-Based Tool for Prediction of Sudden Death in Patients With Non-Ischemic Cardiomyopathy
Acronym: NICMR
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Mayo Clinic (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: WUH 14305; 18-01681 (Other: NYU Langone Institutional Review Board)
Record Dates: First submitted 2015-05-11; First posted 2016-01-18 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Non-ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Whole blood specimens obtained with subject permission, will be retained for the purpose of future genetic research.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an observational study to determine predictors of sudden cardiac death or appropriate ICD therapy in patients with non-ischemic cardiomyopathy. Patients will be followed for 36 months for the occurrence of sudden cardiac death

DETAILED DESCRIPTION:
Non-ischemic cardiomyopathy (NICM) comprises almost one half of the congestive heart failure (CHF) population NICM portends an increased risk for hospitalizations due to CHF as well as death. This population is also at high risk for the occurrence of tachyarrhythmias and has a high incidence of sudden cardiac death (SCD). The risk of SCD can be lowered by the placement of an (intercardioverter defibrillator) ICD. The implantation of an ICD significantly reduces the risk of SCD in patients with NICM and a left ventricular ejection fraction (LVEF) of 35 percent or less. However the implantation of an ICD has short term as well as long term risk associated with it. Many patients receive an ICD who never go on to have appropriate therapy. Current American College of Cardiology/American Heart Association (ACC/AHA) guidelines state that "ICD therapy is recommended for primary prevention of SCD to reduce total mortality in selected patients with nonischemic dilated cardiomyopathy (DCM) or ischemic heart disease at least 40 days post-myocardial infarction(MI) with LVEF of 35% or less and New York Heart Association (NYHA) class II or III symptoms on chronic guideline-directed medical therapy(GDMT), who have reasonable expectation of meaningful survival for more than 1 year." There is a need for new criteria for ICD placement in patients with NICM that are more sensitive and specific than current guidelines.

Delayed enhancement imaging on cardiac magnetic resonance imaging (CMR) has become the gold standard for myocardial scar/necrosis detection. The presence of late gadolinium enhancement (LGE) on CMR which corresponds to myocardial scarring or fibrosis has been shown to be a predictor of adverse outcomes in ischemic cardiomyopathy. There have been few studies evaluating the significance of LGE in patients with NICM, however the results are promising. The presence of LGE has been associated with the incidence of inducible tachycardia by electrophysiology (EP) testing in patients with NICM. LGE has also been associated with an increased risk of morbidity and mortality in a general NICM population.

The investigators plan to enroll patients with NICM with an EF ≤ 40% who have been referred for CMR and follow them for the composite endpoint of sudden cardiac death or an appropriate ICD therapy (Antitachycardic pacing or shock).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed NICM defined as patients whose initial signs or symptoms of cardiomyopathy do not pre-date the time of enrollment for the study by more than six months.
2. LVEF ≤ 40%. (Based on transthoracic echocardiography [Simpson´s Rule])
3. NYHA functional class I-IV
4. Patients aged 18 to 85, both genders and of all races and ethnicities.
5. Patients diagnosed with peripartum cardiomyopathy (PPCM) may be included as long as they are enrolled within six months of initiation of cardiac symptoms.
6. Patients must be competent to give informed consent.

Exclusion Criteria:

1. Significant coronary artery disease > 75% luminal stenosis in at least 1 epicardial vessel, or history of myocardial infarction1 or coronary revascularization.
2. Congenital heart disease.
3. Infiltrative cardiomyopathy (amyloid, sarcoidosis, glycogen storage disease or hemochromatosis).
4. Patients whose heart failure is felt to be secondary to primary valvular disease ( ≥ moderate/severe mitral regurgitation), uncorrected thyroid disease, uncontrolled hypertension despite medical therapy, obstructive or hypertrophic cardiomyopathy, pericardial disease or a systemic illness.
5. Absolute contraindications to undergo CMR (Renal failure with glomerular filtration rate(GFR)<30% or ICD/PPM).
6. Unwilling or unable to provide informed consent.
7. Patients with other life threatening diseases such as malignancy which would likely decrease their life expectancy over the next three years. Any history of malignancy treated with either chest radiation or chemotherapy.
8. Past or present history of alcoholism, or in whose current alcohol consumption exceeds an average of three drinks per day. A past history of cocaine or IV drug abuse as a possible explanation for their cardiomyopathy as well as substance abuse of prescription pain relievers or any illicit drug that may hinder the participant's ability to complete study follow-up.
9. Patients who are post cardiac transplant.
10. Pregnancy.
11. Subjects who are asymptomatic, but are diagnosed with a cardiomyopathy of unknown duration during screening for known familial disease are excluded
12. Patients who are enrolled in other trials with a treatment arm (Patients enrolled in diagnostic trials can be included).
13. Difficulty to attend the follow-up schedule due to a history of medical noncompliance, living a distance from the study center, or anticipated nonresidence in the area for the length of time required for follow-up.
14. Patients on anti-arrhythmics or immunosuppressant drugs.
15. Tachyarrhythmia/Premature Ventricular Contraction (PVC) induced cardiomyopathy which normalizes within 3 months after beginning of treatment of tachyarrhythmia/PVCs.
16. The following patients are excluded for medical reasons: Patients with evidence of chronic liver disease (total bilirubin >3.0mg%) or chronic renal disease (creatinine > or equal to 2.5mg%) are excluded from the study. Subjects who present with an acute worsening of renal function or liver function tests in the setting of worsening heart failure can be enrolled if GFR >30% at the time of CMR.
17. Evidence of ongoing bacteremia or sepsis. Patient with a febrile illness felt to be secondary to myocarditis (even with a non-diagnostic biopsy).
18. Patients who have had a myocardial biopsy that reveals evidence of myocarditis as defined by Dallas criteria or cardiac MRI evidence of myocarditis by Louise criteria are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-ischemic cardiomyopathy and an ejection fraction of ≤40%.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Sudden Cardiac Death or Appropriate ICD Shock Therapy or Anti-tachycardia Pacing or Resuscitated Sudden Cardiac Death | 3 years
  Sudden cardiac death is defined as patients who die suddenly and unexpectedly within 1 hour of cardiac symptoms in the absence of progressive cardiac deterioration, die unexpectedly in bed during sleep and/or die unexpectedly within 24 hours after last being seen alive.
  Appropriate ICD therapy is defined as Shock Therapy or Antitachycardia Pacing.

SECONDARY OUTCOMES:
All cause death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gaztanaga, MD, Principal Investigator — NYU Langone Winthrop University Hospital
Locations (3):
- United States (2):
  - NYU Winthrop Hospital, Mineola, New York
  - Montefiore Medical Center, The Bronx, New York
- University Health Network Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No